CLINICAL TRIAL: NCT04708925
Title: Hypertriglyceridemia-associated Acute Pancreatitis: Apheresis Vs. Conservative Treatment. A Retrospective Study
Brief Title: Hypertriglyceridemia-associated Acute Pancreatitis: Apheresis Vs. Conservative Treatment
Status: Completed | Type: Observational
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, sara dichtwald, Dr, Meir Medical Center
Other Study IDs: 0350-19-MMC
Record Dates: First submitted 2021-01-12; First posted 2021-01-14 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Acute Pancreatitis
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group A- conservative therpay: hypertriglyceridemia-induced acute pancreatitis patients who recieved conservative therapy
- group B- plasmapharesis therapy: hypertriglyceridemia-induced acute pancreatitis patients who recieved plasmapharesis therapy
  Interventions: Other: conservative versus plasmapharesis therapy

INTERVENTIONS:
Other: conservative versus plasmapharesis therapy — conservative versus plasmapharesis therapy
  Groups: group B- plasmapharesis therapy

SUMMARY:
Introduction: Hypertriglyceridemia is one of the etiologies of acute pancreatitis. It may cause severe multi-system disease resulting in high morbidity and mortality. There is controversy regarding the best method to treat it, which includes, among other therapies, high-dose insulin and performing plasma exchange (apheresis).

Aims: Primary outcome - Comparison of 28- day mortality between hypertriglyceridemia-induced acute pancreatitis patients who received conservative therapy versus those who received apheresis therapy. Secondary outcomes: Comparison of morbidity parameters and rate of blood triglycerides level decrease between the groups.

Materials and Methods: A retrospective study based on observational data collection, which will include all patients aged 18--99 who were admitted to the intensive care unit in 2010-2020 in the diagnosis of acute pancreatitis secondary to high blood lipids. Data will be collected from hospital files and computerized systems. Data will include demographics, admission times, ventilation days, pressor support, 28- day mortality,daily triglyceride level, medical history, APACHE-2 score, lactate level, need for dialysis, need for antibiotics and surgical intervention. The study will include 29 patients. All demographic and patient parameters will be statistically examined by a qualified statistician depending on the type of data.

DETAILED DESCRIPTION:
Background: Hypertriglyceridemia causes 1-7% of all acute pancreatitis cases. The mechanism by which excess lipids in the blood cause pancreatitis is not entirely clear. The hypothesis is, that the enzyme lipase, which originates in the pancreas, causes increased breakdown of triglycerides into free fatty acids, which are toxic to endothelial cells and pancreatic acinary cells. In addition, excess fat in the blood increases blood viscosity and impairs blood flow to the pancreas, thus causing necrosis.

There is controversy regarding the best way to treat pancreatitis secondary to hypertriglyceridmia. In addition to fasting, intravenous fluids and analgesia, a number of methods have been used to lower blood lipids, such as heparin and insulin or plasma exchange. Performing plasma exchange causes rapid removal of lipids from the plasma, but it is not yet accepted as the treatment of choice, as there are so far no random prospective studies that have shown an advantage for this treatment method over conservative methods.

The American Society of apheresis defines plasma exchange as a Category 3 indication for the treatment of acute pancreatitis secondary to hyperlipidemia, i.e. as a treatment method whose effectiveness has not been unequivocally proven, and its use is at the discretion of the treating physician.

In the last ten years, the intensive care unit at our institution has treated 29 patients who were admitted due to hypertriglyceridemia induced acute pancreatitis. Some patients were treated conservatively, and some were treated by plasma exchange. We would like to investigate whether there was a difference in mortality rates and morbidity parameters between the groups.

Aims: The primary outcome of this study was to compare 28-days mortality rates among patients who received apheresis versus those who did not. Secondary outcomes were comparison of morbidity parameters between the groups: APACHE score, ICU and hospital length of stay, ventilation days, pressor support, need for renal replacement therapy, need for antibiotics, need for surgical of minimally invasive intervention, and rate of blood triglycerides decrease.

Materials and methods: A retrospective study among patients who were admitted to the ICU between years 2010-2020 due to hypertriglyceridemia-induced acute pancreatitis, a total of 29 cases. Data will be collected from hospital files and computer systems (Chameleon system and iMDsoft software).

Inclusion criteria: All patients aged 18-99 who were admitted to the intensive care unit in Meir medical hospital between years 2010-2020, whose cause of admission was hypertriglyceridemia-induced acute pancreatitis, defined as abdominal pain, elevated levels of amylase and lipase and blood triglyceride level above 1000 mg/dl, without any other apparent etiology of pancreatitis.

Collected data: Patient demographics and medical history including chronic pharmacologic therapy, hospital admission times, ventilation days, inotropic therapy, hemodialysis, daily blood triglyceride level, 28-day mortality, APACHE 2 score, lactate level, antibiotic therapy and need for surgical intervention. All data will be statistically analyzed according to type of data

ELIGIBILITY:
Inclusion Criteria:All patients aged 18-99 who were admitted to the intensive care unit in Meir medical hospital between years 2010-2020, whose cause of admission was hypertriglyceridemia-induced acute pancreatitis, defined as abdominal pain, elevated levels of amylase and lipase and blood triglyceride level above 1000 mg/dl, without any other apparent etiology of pancreatitis.

-

Exclusion Criteria:None

-

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients aged 18-99 who were admitted to the intensive care unit in Meir medical hospital between years 2010-2020, whose cause of admission was hypertriglyceridemia-induced acute pancreatitis, defined as abdominal pain, elevated levels of amylase and lipase and blood triglyceride level above 1000 mg/dl, without any other apparent etiology of pancreatitis.
  -
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
28-day mortality | 28 days
  mortality within 28 days from ICU admission

CONTACTS AND LOCATIONS:
Overall Officials: Sara Dichtwald, MD, Study Chair — Meir Medical Center
Locations (1):
- Meir Medical Center, Kfar Saba, Israel